CLINICAL TRIAL: NCT02343263
Title: Effect of Bupivacaine-infused Fibrin Sealant Application on Post-tonsillectomy Pain & Hemorrhage: a Clinical Trial.
Brief Title: Effect of Bupivacaine-infused Fibrin Sealant Application on Post-tonsillectomy Pain & Hemorrhage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA IND was not obtained
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Bruce Matt, Associate Professor, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1501306006
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative; Postoperative Hemorrhage
Keywords: Tonsillectomy; Adenotonsillectomy; Pain; Hemorrhage
MeSH Terms: conditions — Pain, Postoperative; Postoperative Hemorrhage; Pain; Hemorrhage | interventions — Bupivacaine; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): 44 patients will be randomized to receive no topical treatment to their tonsillectomy (or adenotonsillectomy) wound bed as is the current standard of care at our institution. The wound bed will be treated with instrumentation in the operating room to ensure adequate hemostasis alone.
- Fibrin Sealant Alone (Active Comparator): 44 patients will be randomized to receive application of topical fibrin sealant to their tonsillectomy (or adenotonsillectomy) wound bed to assess the pain reduction benefits of fibrin sealant alone. Prior to application of fibrin sealant, the wound bed will be treated with instrumentation in the operating room to ensure adequate hemostasis.
  Interventions: Biological: Fibrin Sealant
- Bupivacaine-infused Fibrin Sealant (Experimental): 44 patients will be randomized to receive application of topical bupivacaine-infused fibrin sealant to their tonsillectomy (or adenotonsillectomy) wound bed to assess the pain reduction benefits of fibrin sealant alone. Prior to application of fibrin sealant, the wound bed will be treated with instrumentation in the operating room to ensure adequate hemostasis.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 1 milliliter (mL) of 0.75% Bupivacaine Hydrochloride will be infused into 4mL of fibrin sealant (diluting the Bupivacaine HCl to 0.15%). The bupivacaine-infused fibrin sealant will then be applied to the tonsillectomy (or adenotonsillectomy) wound bed.
  Other Names: Marcaine
  Arms: Bupivacaine-infused Fibrin Sealant
Biological: Fibrin Sealant — Fibrin sealant will be applied to the wound bed topically as per product instructions.
  Other Names: Fibrin Glue
  Arms: Fibrin Sealant Alone

SUMMARY:
The purpose of this study is to evaluate the effect of combining two interventions already in use at some institutions for reducing post-operative pain following tonsillectomy or adenotonsillectomy. The standard of care at most institutions is to leave the tonsillectomy wound bed exposed to heal on its own over one to two weeks. At many institutions, surgeons inject or topically apply local anesthetics such as bupivacaine hydrochloride to the tonsillectomy wound bed to help reduce post-operative pain. At other institutions, surgeons apply a layer of fibrin sealant, which is derived from the proteins that help form blood clots in blood, to the tonsillectomy wound bed in order to cover the site and reduce irritation and exposure of the wound bed. Use of fibrin sealant has the additional benefit of potentially reducing postoperative bleeding (hemorrhage) rates. Both the post-tonsillectomy use of bupivacaine (injection and topical) and the use of topical fibrin sealant application have been studied previously in the scientific literature; some studies show a clear benefit, others show no significant reduction in pain when they are used. No studies have documented harm. The purpose of this study is to evaluate the efficacy of infusing bupivacaine anesthetic into the fibrin sealant prior to application to the tonsillectomy wound bed. In this way, the combined product would function as a sort of "medicated bandaid" covering the painful wound bed and slowly delivering an entirely safe total dose of bupivacaine into the wound bed to reduce post-operative pain. Parents will be provided post-operative pain measurements to complete during the first 10 postoperative days and return to the researchers for data analysis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of combining two interventions already in use at some institutions for reducing post-operative pain following tonsillectomy or adenotonsillectomy. The standard of care at most institutions is to leave the tonsillectomy wound bed exposed to heal on its own over one to two weeks. At many institutions, surgeons inject or topically apply local anesthetics such as bupivacaine hydrochloride to the tonsillectomy wound bed to help reduce post-operative pain. At other institutions, surgeons apply a layer of fibrin sealant, which is derived from the proteins that help form blood clots in blood, to the tonsillectomy wound bed in order to cover the site and reduce irritation and exposure of the wound bed. Use of fibrin sealant has the additional benefit of potentially reducing postoperative bleeding (hemorrhage) rates. Both the post-tonsillectomy use of bupivacaine (injection and topical) and the use of topical fibrin sealant application have been studied previously in the scientific literature; some studies show a clear benefit, others show no significant reduction in pain when they are used. No studies have documented harm. The purpose of this study is to evaluate the efficacy of infusing bupivacaine anesthetic into the fibrin sealant prior to application to the tonsillectomy wound bed. In this way, the combined product would function as a sort of "medicated bandaid" covering the painful wound bed and slowly delivering an entirely safe total dose of bupivacaine into the wound bed to reduce post-operative pain.

The hypothesis of this study is that the application of the bupivacaine-infused fibrin sealant will 1) reduce post-operative mean pain scores in children undergoing tonsillectomy or adenotonsillectomy using a validated pediatric pain scoring system, 2) reduce post-operative hemorrhage rates, 3) reduce post-operative vomiting, 4) reduce total doses of post-operative pain medication and narcotic pain medication required, and 5) expedite recovery as determined by return to normal diet and activity level.

The questions specific for this study include: 1) Does bupivacaine-infused fibrin sealant significantly reduce mean postoperative pain scores compared to fibrin sealant alone and compared to leaving the wound bed open to heal?, 2) Does bupivacaine-infused fibrin sealant significantly reduce mean postoperative tonsil hemorrhage rates compared to fibrin sealant alone and compared to leaving the wound bed open to heal? 3) Do children receiving bupivacaine-infused fibrin sealant require less pain medication compared to fibrin sealant alone or to leaving the wound bed open to heal?, 4) Do children receiving bupivacaine-infused fibrin sealant return to normal diet and normal activity sooner compared to fibrin sealant alone or to leaving the wound bed open to heal?, 5) Do the parents of children receiving bupivacaine-infused fibrin sealant make less calls to the clinic or the physician on call compared to fibrin sealant alone or to leaving the wound bed open to heal?

After discussion of the risks and benefits of performing tonsillectomy or adenotonsillectomy per routine, parents will be offered (if child meets inclusion criteria elaborated below) to participate in this research study. This discussion will take place either during the clinic encounter when the patient is signed up for their surgical procedure or on the day of surgery. The Informed Consent Statement will be reviewed with the parent/patient and either the surgical staff, resident investigators, or clinic nursing personnel included in the IRB proposal will be the individuals performing the discussion with the parents. If parents are agreeable to participating in the study and all questions have been asked and no exclusion criteria met, then the child will be enrolled.

The child will be randomized to one of the three treatment arms elaborated in this application. Randomization arms include either: 1) leave wound bed open to heal, 2) application of unaltered fibrin sealant, and 3) application of bupivicaine-induced fibrin sealant. Children will undergo tonsillectomy or adenotonsillectomy per routine, but at the conclusion of the surgical procedure will have either of the 3 treatment options performed as above.

For some children who have clinical concern for sleep disordered breathing or obstructive sleep apnea on a sleep study, the surgical procedure may also involve a direct laryngoscopy and bronchoscopy performed prior to tonsillectomy or adenotonsillectomy. During the laryngoscopy and bronchoscopy, the airway from the level of the mouth to the branches of the windpipe into each lung are inspected with small rigid cameras (endoscopes); if floppiness/collapse (laryngomalacia) of the supraglottis (tissue above the vocal cords) is observed, the child will undergo a laser supraglottoplasty to remove the floppy tissue and relieve the obstruction. If a child has laryngomalacia and supraglottoplasty is performed, the child will then be excluded from the study. Exclusion at this time is based on the creation of an additional wound bed in the throat which could weaken our ability to determine if application of fibrin sealant or bupivacaine-infused fibrin sealant is effective. If during direct laryngoscopy and bronchoscopy, no laryngomalacia is observed and no supraglottoplasty is performed, then the child will continue into the treatment arm into which they were randomized.

After inclusion, randomization, and proceeding with treatment based on the study arm to which the child was randomize, all parents/participants will received standardized post-operative discharge instructions with regard to pain medicine regimens and diet as well as an envelope containing pain assessment questionnaires to be completed 3 times daily for 10 days as a means of documenting pain scores among other data points. The parents will receive a pre-addressed, pre-stamped envelop to facilitate return of their data to the researchers. Currently our clinic nurses call the family of patients approximately 2-3 weeks after surgery to inquire as to how the child is doing and to ensure that if the family desires a follow up appointment that one will be made. Parents of children included in this study will receive a similar phone call during the same approximate time frame either by the clinic nurses or by the surgical staff or resident investigators, but additional specific questions regarding post-operative bleeding and pain control will be documented for research purposes. Additionally, during this phone call, parents will be reminded to complete and return their post-operative pain assessment sheets in the provided pre-addressed, pre-stamped envelopes they received on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. All children aged 1 through age 12 and weighing >10 kilograms who are scheduled for tonsillectomy or adenotonsillectomy for the following indications by surgical staff included in the IRB submission will be considered for inclusion in the study.

A) Chronic Pharyngitis / Recurrent Tonsillitis B) PAPFA (Periodic Aphthous Ulcers / Pharyngitis / Fevers / Adenopathy) Syndrome C) Upper Aerodigestive Obstruction Symptoms felt to be related to tonsil size. D) Adenotonsillar Hypertrophy (enlarged tonsils and adenoids) E) Obstructive Sleep Apnea (clinical diagnosis or by Polysomnogram [sleep study]) F) Chronic/Recurrent Tonsillolithiasis (tonsil stones)

Exclusion Criteria:

1. Undergoing additional surgical procedures within 14 days preceding or following the tonsillectomy or adenotonsillectomy which could affect pain assessment scores.
2. Additional concurrent surgical procedures (other than direct laryngoscopy, bronchoscopy, nasal endoscopy, ear examination under anesthesia, cerumen removal, or myringotomy with ear ventilation tube placement)

2. If decision is made to perform supraglottoplasty for laryngomalacia intraoperatively

3. Tonsillectomy or adenotonsillectomy for concern of malignancy of unknown primary

4. Documented aprotinin allergy

5. Documented amide anesthetic allergy

6. Documented bleeding disorder

7. Documented anticoagulant use

8. Documented chronic pain disorder

9. Documented chronic use of prescription narcotics or methadone

10. Documented history of substance abuse or illicit drug use

11. Documented history of alcoholism or alcohol abuse

12. Gastrostomy/orogastric/nasogastric tube placement/use

13. Planned postoperative ICU placement

14. Refusal to participate

15. Exclusion at judgment of investigator (Language barriers, Ward of Court, etc.)

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H Matt, MD,MSc, Principal Investigator — Indiana University
Locations (1):
- Riley Childrens' Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed due for administrative reasons
Pre-assignment Details: Study closed due for administrative reasons. Subjects fell out of study due to a number of reasons, including receiving a laser supraglottoplasty which was an exclusion criteria. Also, failure to complete study. Also our IRB later required a FDA IND which we did not obtain, so study was stopped
Groups:
- Control Arm: Control Arm did not receive any Fibrin sealant nor Bupivacaine
- Fibrin Sealant Alone: Fibrin Sealant Alone- subjects received only fibrin sealant to tonsillar fossa
- Bupivacaine-infused Fibrin Sealant: Bupivacaine-infused Fibrin Sealant was placed in tonsillar fossa of subjects
Period: Overall Study
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Started | 5 (Study closed due for administrative reasons) | 3 | 1
Completed (Study closed due for administrative reasons) | 0 (Study closed due for administrative reasons) | 0 | 0
Not Completed | 5 | 3 | 1
Not completed — Physician Decision | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Population: study terminated due to FDA requirement for a investigational new drug application requirement
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant | Total
Number analyzed (Participants) | 5 | 3 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 1 | 9
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (1.8) | 3.7 (2.9) | 8 (0) | 5.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 4 | 2 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 1 | 9
study closed for administrative reasons [Count of Participants; unit: Participants] | 5 | 3 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Hemorrhage; Study Terminated Due to FDA Requirement for a Investigational New Drug Application Requirement
Description: Tonsillectomy (and adenotonsillectomy) are associated with a 3-5% postoperative hemorrhage risk from the tonsillectomy wound beds across the United States; our institution has a calculated average of between 4% - 5%. Parents will be contacted 2 to 3 weeks following their procedure and inquiries about post-operative bleeding will be made. Bleeding >1 tablespoon or that requires A) presentation to an emergency department, B) admission to a hospital, or C) return to the operating room will be considered significant post-operative hemorrhage. Distinction will also be made between early (<24 hours after surgery) and late (>24 hours after surgery) postoperative bleeding. The bleeding risk after 2 weeks from surgery is exceedingly small. No prior studies have identified any increased risk with utilizing either fibrin sealant or bupivacaine. This study will evaluate whether the intervention reduces bleeding risk.
Time Frame: 14 days
Population: Data not collected
Groups:
- Control Arm: study terminated due to FDA requirement for a investigational new drug application requirement. Subjects did not receive Fibrin sealant nor Bupivacaine
- Fibrin Sealant Alone: subjects received fibrin sealant to tonsillar fossa
- Bupivacaine-infused Fibrin Sealant: subjects received Bupivacaine-infused Fibrin Sealant to tonsillar fossa
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Postoperative Pain; Study Terminated Due to FDA Requirement for a Investigational New Drug Application Requirement
Description: Parents/caregivers will be asked to perform thrice daily pain assessments utilizing a validated postoperative pain measurement scale for the 10 days after surgery. study terminated due to FDA requirement for a investigational new drug application requirement
Time Frame: 10 days
Population: data not collected
Groups:
- Control Arm: subjects did not receive fibrin sealant nor bupivacaine
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Total Pain Medication Usage
Description: The postoperative pain assessment sheets will contain a daily entry for the estimated total doses of pain medication required and will distinguish between the need for narcotic and non-narcotic pain medication requirements.
Time Frame: 10 days
Population: data not collected
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Return to Normal Diet
Description: The postoperative pain assessment sheets will contain a daily entry for the estimated number of postoperative days until patient returned to normal diet.
Time Frame: 10 days
Population: data not collected
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Required Calls to Healthcare Personnel (Either the Clinic or the Physician on Call Overnight)
Description: The postoperative pain assessment sheets will contain a daily entry for the estimated number of required calls to the clinic or to the physician on call overnight.
Time Frame: 10 days
Population: data not collected
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Postoperative Nausea & Emesis
Description: The postoperative pain assessment sheets will contain a daily entry for the estimated number of episodes of vomiting the patient experienced.
Time Frame: 10 days
Population: data not collected
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Time to Return to Normal Activity
Description: The postoperative pain assessment sheets will contain a daily entry for the estimated number of postoperative days until patient returned to normal activity level.
Time Frame: 10 days
Population: data not collected
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse events not monitored
Description: adverse events not monitored
Groups:
- Fibrin Sealant Alone: subjects received fibrin sealant alone to the tonsillar fossa
- Bupivacaine-infused Fibrin Sealant: subjects received Bupivacaine-infused Fibrin Sealant to the tonsillar fossa
Arm/Group | Control Arm | Fibrin Sealant Alone | Bupivacaine-infused Fibrin Sealant
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
study closed due to need for FDA investigational new drug application.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02343263/Prot_SAP_000.pdf